CLINICAL TRIAL: NCT01141946
Title: Pleural Ultrasonography in Lung Cancer - PULC
Brief Title: Pleural Ultrasonography in Lung Cancer
Acronym: CT0018
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government); Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other); Society of University Surgeons (Other)
Responsible Party: Sponsor
Other Study IDs: CE 10.046
Record Dates: First submitted 2010-06-07; First posted 2010-06-11 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2011-06

CONDITIONS: Lung Cancer
Keywords: lung cancer; pleural effusion; post-op care; diaphragmatic ultrasound
MeSH Terms: conditions — Lung Neoplasms; Pleural Effusion | interventions — Thoracentesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: thoracic ultrasound — All patients will receive pre-operative pleural-based ultrasound during their initial consultation.
Procedure: pleural aspiration — Before proceeding to pleural aspiration, a radiography of the chest will be performed in order to ascertain the presence of a pleural effusion.

SUMMARY:
Lung cancer remains the leading cause of mortality from malignant diseases in both men and women worldwide. Accurate diagnosis, staging and therapeutic targeting of lung cancer and other pulmonary pathology are vital with regards to providing patients with expedient and accurate treatment and treatment plans. The pre-operative evaluation and consultation in patients who are to undergo operative staging or resection for lung cancer is multidimensional and involves detailed history taking, physical examination and review of imaging studies. Two important elements of both staging and pre-operative evaluation include the evaluation of: (1) the pleural space for malignant pleural effusion and (2) the diaphragm for appropriate movement. At this point in time, the pleural space evaluation is being performed using CT scan which does not allow the acquisition of real-time cytological material from pleural effusions due to the fact that the CT scans are done in a diagnostic setting. Diaphragmatic movement/excursion is not currently being assessed pre-operatively and its impact on staging and post-operative pulmonary function is unknown.

Malignant pleural effusion is recognized as a poor prognosticator in non-small cell lung cancer patients and has recently been upgraded from a T4 to an M1a status in the new edition of the AJCC NSCLC Staging System (7th Edition). The appreciation of the poor prognosis related to malignant effusion has upgraded the stage from a Stage IIIb to a stage IV. Recognizing the stage early allows for more precise prognostication of disease and can lead to precision and streamlining of treatment plans for thoracic surgeons and oncologists.

DETAILED DESCRIPTION:
Hypotheses:

1. Pleural ultrasonography with evaluation, quantification and aspiration of pleural effusion allows for improved pre-operative staging and alters decision-making patterns for lung cancer patients.
2. Pleural ultrasonography with evaluation of appropriate diaphragmatic respiratory movement can predict post-operative complications in patient undergoing lung cancer surgery.

Objectives:

The goals of this project within the program are to:

1. Evaluate the improvement in pre-operative staging with the addition of pre-operative pleural ultrasonography for malignant pleural effusion.
2. Evaluate the ability of pre-operative diaphragmatic ultrasound to predict post-operative morbidity following pulmonary surgery.

Methodology:

This study will consist of a prospective evaluation of surgeon-performed pleural and diaphragmatic ultrasound in the pre-operative evaluation of lung cancer patients. All patients being seen in the thoracic surgery pre-operative clinic with the new or presumed diagnosis of lung cancer will be approached for prospective enrolment into the study. Consented patients will undergo standard history and physical examination by the treating thoracic surgeon. During or after the physical examination, PULC will be performed by the study investigators.

Measurements will include: (1) bilateral diaphragmatic excursion during sniffing, (2) pleural fluid evaluation in bilateral costophrenic sulci. Should pleural fluid be found on the ipsilateral side to the mass (tumor), the fluid will be aspirated under sterile conditions in the clinic and sent for cytology analysis. US evaluation will be performed in the upright, supine and decubitus position.

Results will be analyzed using parametric methodology in order to ascertain the additional information gained and the change in staging (upstaging) with the addition of PULC to standard history and physical examination during the initial evaluation of thoracic surgical patients.

The study will enrol 50 patients. Recruitment will occur at the thoracic outpatient surgical clinic at the CHUM. Enrolment is expected at a level of five patients per week and therefore the study recruitment is expected to take 2.5 months.

Impact:

The potential impact of a positive trial will change the way clinicians evaluate, stage and risk stratify patients who are to undergo operative interventions for lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Lung lesion being evaluated for surgery during initial consultation with a thoracic surgeon

Exclusion Criteria:

* Age < 18 years old
* Inability to consent for the study
* Chest wall anatomy precluding PULC
* Inability to sit upright
* Medications including Warfarin (Coumadin) or Clopidogrel (Plavix) in patient requiring pleural fluid aspiration
* Active cutaneous infection overlying proposed puncture site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The improvement in pre-operative staging with the addition of pre-operative pleural ultrasonography for malignant pleural effusion. | 3 months

SECONDARY OUTCOMES:
The ability of pre-operative diaphragmatic ultrasound to predict post-operative morbidity following pulmonary surgery. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Moishe Liberman, MD, PhD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada